CLINICAL TRIAL: NCT00878215
Title: Clinical Application of Image-Guided Liver Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The image-guidance system became commercially available
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201104308
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Results first posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-01

CONDITIONS: Hepatocellular Cancer
Keywords: Image Guided Liver Surgery
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Phase 1:Localize Anatomical Points on Liver Surface (Experimental): -The surgeon will use image-guided surgery equipment to create the mapping with 3-D pictures of the participants liver. Laser range scanning will also be used to take 3-D pictures of the liver surface. The participant will then have planned standard surgery.
  Interventions: Device: Explorer Liver Image Guided System; Device: Explorer Liver Passive Tracking; Procedure: Liver surgery
- Phase 2: Ceramic bead (Experimental): -The surgeon will use image-guided surgery to create the mapping with 3-D pictures of the liver. During the surgery, a ceramic bead will be placed in a pre-operatively determined target location within the tumor using image-guided surgery. Standard surgical procedures will then be used to remove the tumors. Magnetic resonance (MR) images of the resected liver will confirm targeting accuracy.
  Interventions: Device: Explorer Liver Image Guided System; Device: Explorer Liver Passive Tracking; Procedure: Liver surgery
- Phase 3: Ablative therapy (Experimental): -The surgeon will use image-guided surgery to create the mapping with 3-D pictures of the liver. The liver tumors will be ablated using image-guided surgery. Standard surgical procedures will then be used to remove the portion of the liver that has the ablated tumors. The accuracy of the ablation will be confirmed via pathology sectioning.
  Interventions: Device: Explorer Liver Image Guided System; Device: Explorer Liver Passive Tracking; Procedure: Liver surgery; Procedure: Liver abalation
- Phase 4: Ablative therapy (not liver resection candidates) (Experimental): -This phase is for patients who otherwise do not qualify to have a portion of their liver to be surgically removed. The surgeon will use image-guidance to create the mapping with 3-D pictures of the liver. The tumors will be ablated using image-guided therapy.
  Interventions: Device: Explorer Liver Image Guided System; Device: Explorer Liver Passive Tracking; Procedure: Liver abalation

INTERVENTIONS:
Device: Explorer Liver Image Guided System
Device: Explorer Liver Passive Tracking
Procedure: Liver surgery — -Standard of care
  Arms: Phase 1:Localize Anatomical Points on Liver Surface; Phase 2: Ceramic bead; Phase 3: Ablative therapy
Procedure: Liver abalation — -Standard of care
  Arms: Phase 3: Ablative therapy; Phase 4: Ablative therapy (not liver resection candidates)

SUMMARY:
Image-guided surgery is a new technology, which is used to create 3-D pictures that generate a map of the liver. This map will allow surgeons to know the exact anatomical location of their instruments, including instances when direct visualization is not possible. This study is designed to determine the safety and feasibility of using image-guided techniques for treatment of liver tumors. The overall goal of this study is to use image-guided surgery for the improvement of the surgeon's ability to remove liver tumors.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained.
* Patient must be 18 years or older.
* Are male or non-pregnant, non-lactating females. Liver resection or ablation could be harmful to an unborn child therefore, is not recommended during pregnancy. After informed consent is obtained, women of childbearing potential will be required to have a blood or urine pregnancy test. All consented patients of childbearing potential will be advised to use adequate birth control (oral, implanted, or barrier methods) along with their sexual partners while being considered for liver tumor resection or ablation and at least up to a month following surgery.
* Patients enrolled in Phase I must be candidates for surgical liver resection per a treating surgeon's discretion. Patients enrolled in Phase 2-3 must be candidates for surgical liver resection of liver mass. Patients enrolled in Phase 4 must be candidates for surgical ablation, but not candidates for surgical resection.
* Patients are scheduled clinically for use of the Pathfinder Explorer Liver Image Guided System which is indicated for open liver surgical procedures where image-guidance may be appropriate and where the patient can tolerate long apneic periods under general anesthesia.

Exclusion Criteria:

* Any condition which, in the judgment of the investigator, might increase the risk to the subject or decrease the chance of obtaining satisfactory data to achieve the objectives of the study.
* Mental condition rendering the subject or his/her legal representative unable to understand informed consent to the nature, scope, and possible consequences of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2002-10-24 (Actual); Primary Completion 2011-05-25 (Actual); Study Completion 2011-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William C Chapman, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosen CB. Management of Hepatic Metastases. Cancer Control. 1998 May;5(3 Suppl 1):30-31. doi: 10.1177/107327489800503S11. No abstract available. PMID 10762479
- [Background] Sardi A, Akbarov A, Conaway G. Management of primary and metastatic tumors to the liver. Oncology (Williston Park). 1996 Jun;10(6):911-25; discussion 926, 929-30. PMID 8823803
- [Background] Dick EA, Taylor-Robinson SD, Thomas HC, Gedroyc WM. Ablative therapy for liver tumours. Gut. 2002 May;50(5):733-9. doi: 10.1136/gut.50.5.733. PMID 11950826
- [Background] Parikh AA, Curley SA, Fornage BD, Ellis LM. Radiofrequency ablation of hepatic metastases. Semin Oncol. 2002 Apr;29(2):168-82. doi: 10.1053/sonc.2002.31673. PMID 11951215
- [Background] Arun KS, Huang TS, Blostein SD. Least-squares fitting of two 3-d point sets. IEEE Trans Pattern Anal Mach Intell. 1987 May;9(5):698-700. doi: 10.1109/tpami.1987.4767965. PMID 21869429
- [Background] Horn BKP.closed-form solution of absolute orientation using unit quaternions 4:629-642,1987
- [Background] Besl PM,McKay ND.A method for registraion of 3-D shapes.IEEE Transaactions on Pattern Analysis and Machine Intelligence 14:239-256,1992
- [Background] Cash DM,Siha Tk,Chapman,WC.Fast, accurate surface acquistion using a laser range scanner for image-guided surgical system.SPIE Medical Imaging,2002
- [Background] Stefansic JD, Bass WA, Hartmann SL, Beasley RA, Sinha TK, Cash DM, Herline AJ, Galloway RL Jr. Design and implementation of a PC-based image-guided surgical system. Comput Methods Programs Biomed. 2002 Nov;69(3):211-24. doi: 10.1016/s0169-2607(01)00192-4. PMID 12204449
- [Background] Herline AJ, Stefansic JD, Debelak JP, Hartmann SL, Pinson CW, Galloway RL, Chapman WC. Image-guided surgery: preliminary feasibility studies of frameless stereotactic liver surgery. Arch Surg. 1999 Jun;134(6):644-9; discussion 649-50. doi: 10.1001/archsurg.134.6.644. PMID 10367875
- [Background] Herline AJ, Herring JL, Stefansic JD, Chapman WC, Galloway RL Jr, Dawant BM. Surface registration for use in interactive, image-guided liver surgery. Comput Aided Surg. 2000;5(1):11-7. doi: 10.1002/(SICI)1097-0150(2000)5:13.0.CO;2-G. PMID 10767091
- [Background] Pan S,Dawant BM.Automatic 3-D segmentation of the liver from abdominal CT images: a level-set approach. Proceedings of SPIE 4322:128-138,2001.
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 10/24/2002 with the first participant enrolled on 12/27/2002 and the final participant was enrolled on 05/25/2011.
Period: Overall Study
Arm/Group | Phase 1:Localize Anatomical Points on Liver Surface | Phase 2: Ceramic Bead | Phase 3: Ablative Therapy | Phase 4: Ablative Therapy (Not Liver Resection Candidates)
Started | 21 | 19 | 0 (Phase 3 not performed because the liver imaging system became commercially available) | 0 (Phase 4 not performed because the liver imaging system became commercially available)
Completed | 21 | 9 | 0 | 0
Not Completed | 0 | 10 | 0 | 0
Not completed — Determined to be ineligible | 0 | 10 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1:Localize Anatomical Points on Liver Surface | Phase 2: Ceramic Bead | Phase 3: Ablative Therapy | Phase 4: Ablative Therapy (Not Liver Resection Candidates) | Total
Number analyzed (Participants) | 21 | 19 | 0 | 0 | 40
Age, Continuous [Median (Full Range); unit: years] | 60 [36 to 81] | 58 [25 to 78] |  |  | 59 [25 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 14 |  |  | 20
  Male | 15 | 5 |  |  | 20
Region of Enrollment [Number; unit: participants]
  United States | 21 | 19 |  |  | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Have a Successful Intraoperative Registrations (Phase 1 Portion of Study)
Description: * 10 successful intraoperative registrations with no more than 30% failure rate over all the cases will be considered a successful endpoint
  * A successful registration is defined as one which yields an RMS surface residual of ≤ 10 mm and is determined to be success after qualitative evaluation.
Time Frame: Completion of surgery
Population: 2 patients were excluded due to the fact that liver surface data was not acquired for these cases due to equipment malfunctions and not due to a failure in the guidance method in general.
Measure: Number; unit: participants
Arm/Group | Phase 1:Localize Anatomical Points on Liver Surface
Number analyzed (Participants) | 19
participants | 18

2. Primary Outcome: Accuracy With Which Image-guided Surgery (IGS) Can be Used to Implant a Ceramic Bead Inside a Tumor as Measured by Successful Deliveries of the Bead to Within 8mm of the Pre-operatively Planned Target Point (Phase 2 Portion of Study)
Description: * Calculation of bead delivery accuracy using the IGS system involves the acquisition of images of the resected specimen and then the co-registration of the post-resection images to the pre-operative image set. Given that the target location is marked in the pre-operative image set and the registration calculation allows an overlay of the two image sets a Euclidean distance error can be calculated between the true bead location and the pre-operatively determined target. Given that the error involved in computing the registration between the two image sets is included within the bead delivery target error calculation it is imperative that the impact of registration error is minimized.
  * Numbers represented are the distance between the planned target site and the true bead location
Time Frame: Completion of surgery
Population: 10 patients were excluded as they were determined to be ineligible after enrollment but prior to surgery.
Measure: Number; unit: mm
Arm/Group | Phase 2: Ceramic Bead
Number analyzed (Participants) | 9
mm
  Case 1 | 17.3
  Case 2 | 16.6
  Case 3 | 4.6
  Case 4 | 15.9
  Case 5 | 8.8
  Case 6 | 10.9
  Case 7 | 4.7
  Case 8 | 13.0
  Case 9 | 25.6

3. Primary Outcome: Target Accuracy of an Ablation Probe Using Image-guided Surgery Technology as Measured by the Number of Participants Who Had Ablation Burns Within a 5mm Radius of the Tumor Centroid (Phase 3 Portion of Study)
Description: -A measurement of the ablation probe placement via the burn zone will be performed by pathology via specimen sectioning.
Time Frame: Completion of surgery
Population: The study closed early as the imaging-guidance system became commercially available as the Explorer Liver Image Guided System and the Explorer Liver Passive Tracking device.
Arm/Group | Phase 3: Ablative Therapy
Number analyzed (Participants) | 0

4. Primary Outcome: The Number of Participants Who Have Complete Ablation According to Early Post-ablative Imaging Studies as Well as no Recurrence of the Tumor Within 6 Months (Phase 4 Portion of the Study)
Description: -A successful endpoint will be a 90% success rate of complete ablation according to early post-ablative imaging studies as well as no recurrence of the tumor within 6 months.
Time Frame: 6 months post-ablation
Population: as for outcome 3
Arm/Group | Phase 4: Ablative Therapy (Not Liver Resection Candidates)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Phase 1:Localize Anatomical Points on Liver Surface | Phase 2: Ceramic Bead | Phase 3: Ablative Therapy | Phase 4: Ablative Therapy (Not Liver Resection Candidates)
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/21 | 0/19 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No